CLINICAL TRIAL: NCT05281016
Title: Integrating Community LITE Programme Into a School-clinic-community Partnership as an Online Family-based Intervention to Combat Childhood Obesity
Brief Title: Integrating Community LITE Programme as an Online Family-based Intervention to Combat Childhood Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Duke University (Other); Sport Singapore (Unknown); Health Promotion Board, Singapore (Other Government); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20210006
Record Dates: First submitted 2022-03-06; First posted 2022-03-15 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Pediatric Obesity
Keywords: child health; Body Mass Index; Healthy Lifestyle; Community Networks; internet-based intervention; Diet, Food, and Nutrition; Parenting
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Intervention Control Group (Experimental): Participants randomised to the Control Group will be offered standard care and will be introduced to 6 month delayed intervention which consists of the online community LITE programme.
  Interventions: Behavioral: Usual Care; Behavioral: Online community LITE programme
- Intervention Group (Experimental): Participants randomised to the Intervention Group will receive standard care plus invitation to participate in the online community LITE programme for 4-5 months.
  Interventions: Behavioral: Usual Care; Behavioral: Online community LITE programme

INTERVENTIONS:
Behavioral: Usual Care — Participants will be offered standard care which consists of the following:
  * Clinic consultation with physician and dietician,
  * pamphlets on weight management principles.
Behavioral: Online community LITE programme — Participants will be invited to participate in the online community LITE programme. Participants will also receive basic sports equipment for the online programme.
  The online community LITE programme will consist of 2 sessions a week for 4-5 months. Each session is 1 hour long. The programme will deliver 3 domains: physical activity, nutrition and behaviour. It consists of relatively unstructured sessions comprising of cooking and nutrition classes, games and sports and peer support.

SUMMARY:
Childhood obesity in Singapore is rising with a record prevalence of 13% in 2017 (1). Given that 70% of overweight children remain so into adulthood (2), this will further increase the public health epidemic of diabetes among Singaporeans. Early intervention is thus critical to improve the weight trajectory of overweight children and foster life long healthy lifestyle habits. Family-based interventions combining dietary, physical activity and behavioural interventions are currently recommended as the best practice in the management of childhood obesity in children younger than 12 years old (3-7). Our pilot study on family-based intervention in the tertiary setting demonstrated feasibility and short-term effectiveness. However, its outreach and sustainable results are limited. Currently, school-based screening, weight management clinics and community recreational facilities are operating in silos with limited effectiveness. Here, the investigators will integrate our family-based intervention into a school, clinic and community partnership to achieve an impactful and sustainable outcome for families with overweight children.

The community Lifestyle InTervention for Everyone (LITE) program is a structured, group family-based multicomponent lifestyle intervention. Community LITE program will introduce various exercise programs within the family based online sessions to reduce perceived barrier and promote self-efficacy of community sports facilities to increase physical activity. Children have minimal control over their food and physical activity choices especially in current obesogenic environment (8). Parents are the most important influencers(9) to impose interventions for childhood obesity through parental practices and parenting style(10). Therefore, they are the main focus of the community-based intervention program.

DETAILED DESCRIPTION:
The investigators hypothesize that our community LITE program can reduce the prevalence of overweight children aged 6-12 years old in Singapore with sustainable lasting effects by encouraging healthy lifestyle and behaviours. The investigators will test our hypothesis with the following aims:

Primary aim: To investigate whether community LITE programme will lead to a reduction in Body Mass Index (BMI) z-score. Intervention outcome will be compared with that from the usual care at 6 months and 12 months.

Secondary aims:

1. To demonstrate implementation feasibility and acceptability of the community LITE programme
2. To estimate cost and cost effectiveness of programme
3. To estimate the effectiveness of programme. Children will demonstrate improvements in health outcomes at 6-months and 12 months, including waist-height, blood pressure, fruits and vegetables intake and MVPA level at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Overweight as defined by BMI percentile of above 90th percentile
* Age 6- 12 years old
* Ability to provide informed consent

Exclusion Criteria:

* Patients with secondary causes of obesity especially genetic syndromes e.g. Trisomy 21, Prader-Willi, and those who are taking medications that can affect weight status.
* Intellectual disability, poor level of spoken English (including their parent/carer)
* Significant medical illness that precludes physical activity and significant psychiatric illness
* Sibling who is already participating in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) | Baseline, 6 months and 12 months
  Measure the change in BMI at baseline, 6 months and 12 months. Body mass index (BMI) will be calculated as kg/m2

SECONDARY OUTCOMES:
Change in waist circumference | Baseline, 6 months and 12 months
  Measure change in waist circumference at baseline, 6 months and 12 months. Waist circumference is measured at the narrowest point between the lower costal (rib) border and the iliac crest using a non-extensible steel tape.
Change in blood pressure | Baseline, 6 months and 12 months
  Measure change in blood pressure at baseline, 6 months and 12 months. Blood pressure will be measured in mmHg via an electronic sphygmomanometer. Both systolic and diastolic blood pressure will be measured.
Change in servings of fruits and vegetables | Baseline, 6 months and 12 months
  Measure change in number of servings of fruits and vegetables using food frequency questionnaire at baseline, 6 months and 12 months .
Change in physical activity | Baseline, 6 months and 12 months
  Measure change in physical activity using results from accelerometer to assess time spent on sedentary and moderate to vigorous physical activity at baseline, 6 months and 12 months.
Change in quality of life | Baseline, 6 months and 12 months
  Measure change in quality of life at baseline, 6 months and 12 months using the Pediatric Quality of Life Inventory (PedsQL; Singapore version 4). PedsQL is a comprehensive and multi-dimensional construct that includes physical, emotional, and social functioning to assess quality of life in the children. It uses a 5-point Likert scale where 0= never, 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always. Items will be reverse scored and linearly transformed to a 0-100 scale so that higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Chu Shan Chew, MBBS, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers based on the informed consent form